CLINICAL TRIAL: NCT01688128
Title: An Open-label, Controlled, Cross-over Trial of Ubiquitous SR-based Memory Advancement and Rehabilitation Training (U-SMART) in Mild Cognitive Impairment
Brief Title: Efficacy of Ubiquitous SR-based Memory Advancement and Rehabilitation Training (U-SMART)
Acronym: U-SMART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: KT Corporation (Industry)
Responsible Party: Principal Investigator, Ki Woong Kim, Professor, department of neuropsychiatry, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E-1207/162-001
Record Dates: First submitted 2012-09-12; First posted 2012-09-19 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive impairment; Cognitive rehabilitation; Cognitive therapy; Spaced retrieval Training; Alzheimer's disease; Memory enhancement; U-healthcare
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention_Control group (Experimental): Phase I: U-SMART for 4 weeks (2 session/week); Washout: for 2 weeks; Phase II: No intervention for 4 weeks
  Interventions: Device: Phase I U-SMART (4 wks); Other: Washout (2 wks)
- Control_Intervention group (Experimental): Phase I: No intervention for 4 weeks; Washout: for 2 weeks; Phase II: U-SMART for 4 weeks (2 session/week)
  Interventions: Other: Washout (2 wks); Device: Phase II U-SMART (4 wks)

INTERVENTIONS:
Device: Phase I U-SMART (4 wks) — Intervention_Control Group, 4-weeks U-SMART(2 session/week); Control_Intervention Group, no intervention
  Arms: Intervention_Control group
Other: Washout (2 wks) — 2-weeks wash out period in both arms
Device: Phase II U-SMART (4 wks) — Intervention_Control Group, no intervention; Control_Intervention Group, 4-weeks U-SMART(2 session/week, Crossover design)
  Arms: Control_Intervention group

SUMMARY:
The purpose of this study is to examine the efficacy of the Ubiquitous Spaced Retrieval-based Memory Advancement and Rehabilitation Training (U-SMART) in the elderly individuals with mild cognitive impairment (MCI) by an open-label, controlled, crossover Trial.

DETAILED DESCRIPTION:
The Spaced Retrieval-based Memory Advancement and Rehabilitation Training (SMART) which consisted of 24 one-hour face-to-face sessions (Lee, Park et al. 2009) was developed based on the spaced retrieval training (SRT), which was effective in improving memory retention span of very mild to mild Alzheimer's disease patients. The Ubiquitous SMART (U-SMART) by transforming the current SMART to a self-administered program using an application working on IPAD was developed, and showed its feasibility and efficacy in the elderly individuals with mild cognitive impairment in the preliminary study. (ClinicalTrials.gov ID: NCT01628653) To validate the efficacy of the U-SMART, an open-label, controlled, crossover design of clinical trial were planned in this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55-90
* Educational level above 1 year and confirmed literacy
* Diagnosed to mild cognitive impairment by International Working Group on Mild Cognitive Impairment
* Clinical Dementia Rating (CDR) of 0 or 0.5

Exclusion Criteria:

* Diagnosed to dementia by DSM-IV
* Evidence of delirium, confusion
* Any neurological conditions causing cognitive decline such as Parkinson's disease, brain hemorrhage, brain tumor, normal pressure hydrocephalus
* Evidence of severe cerebrovascular pathology
* History of loss-of-consciousness over 1 hour due to head trauma or repetitive head trauma of mild severity
* History of substance abuse or dependence such as alcohol
* Presence of depressive symptoms that could influence cognitive function
* Presence of medical comorbidities that could result in cognitive decline Use of medication that could influence cognitive function seriously

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in the Word List Test (memory, recall, recognition) of the CERAD Neuropsychological Assessment Battery before and after phase I intervention and before and after phase II intervention (crossover part of the study) | Baseline, 5 weeks, 11weeks
  To evaluate the efficacy of the U-SMART, the Word List Memory Test (WLMT), Word List Recall Test (WLRT), Word List Recognition Test (WLRcT) of the CERAD neuropsychological assessment battery were applied to all participants.

SECONDARY OUTCOMES:
Change in the Subjective Memory Complaints Questionnaire (SMCQ) before and after phase I intervention and before and after phase II intervention (crossover part of the study) | Baseline, 5 weeks, 11weeks
  To evaluate the subjective memory improvement after the U-SMART, the Subjective Memory Complaints Questionnaire(SMCQ) was applied to all participants.
Change in the Geriatric Depression Scale (GDS) before and after phase I intervention and before and after phase II intervention (crossover part of the study) | Baseline, 5 weeks, 11weeks
  To evaluate the subjective mood after the U-SMART, the Geriatric Depression Scale was applied to all participants.
Change in the Mini-Mental State Examination before and after phase I intervention and before and after phase II intervention (crossover part of the study) | Baseline, 5 weeks, 11weeks
  To evaluate the global cognitive function after the U-SMART, the Mini-Mental State Examination was applied to all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Woong Kim, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital, Seong-nam, Korea
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Han JW, Son KL, Byun HJ, Ko JW, Kim K, Hong JW, Kim TH, Kim KW. Efficacy of the Ubiquitous Spaced Retrieval-based Memory Advancement and Rehabilitation Training (USMART) program among patients with mild cognitive impairment: a randomized controlled crossover trial. Alzheimers Res Ther. 2017 Jun 6;9(1):39. doi: 10.1186/s13195-017-0264-8. PMID 28587629